CLINICAL TRIAL: NCT05928611
Title: Effect of Intraligmentary Dexamethasone on Anesthetic Efficacy of Inferior Alveolar Nerve Block Versus Buccal Infiltratation in Lower First Molars With Irreversible Pulpitis and Apical Periodontits: A Randomized Clinical Trial
Brief Title: Intraligmentary Dexamethasone in Lower First Molars With Irreversible Pulpitis and Apical Periodontits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wafaa Rezk Elshafaey, Prof.Dr. Angie Galal Ghoneim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDO 3 - 3 - 5
Record Dates: First submitted 2023-06-15; First posted 2023-07-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pulpitis - Irreversible
Keywords: " irreversible pulpitis with apical periodontitis"
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inferior alveolar nerve block (Active Comparator): Using 1.8ml of 4% articaine HCL 1:100,000 epinehrine
  Interventions: Procedure: Inferior alveolar nerve block
- Inferior alveolar nerve block with intraligmentary dexamethasone (Experimental): Using 1.8ml of 4% articaine HCL 1:100,000 epinehrine for inferior alveolar nerve block and 0.4 mL of 8 mg/ 2mLdexamethasone for intraligmentary injection
  Interventions: Procedure: Inferior alveolar nerve block with dexamethasone
- Buccal infiltratation with intraligmentary dexamethasone (Experimental): Using 1.8ml of 4% articaine HCL 1:100,000 epinehrine for buccal infiltratation and 0.4 mL of 8 mg/ 2mLdexamethasone for intraligmentary injection
  Interventions: Procedure: Buccal infiltratation with dexamethasone

INTERVENTIONS:
Procedure: Inferior alveolar nerve block with dexamethasone — Using articaine for inferior alveolar block with intraligmentary dexamethasone
  Arms: Inferior alveolar nerve block with intraligmentary dexamethasone
Procedure: Buccal infiltratation with dexamethasone — Using articaine for buccal infiltratation with intraligmentary dexamethasone
  Arms: Buccal infiltratation with intraligmentary dexamethasone
Procedure: Inferior alveolar nerve block — Using articaine for injection
  Arms: Inferior alveolar nerve block

SUMMARY:
Using intraligmentary dexamethasone to reduce the pain intensity during and after root canal preparation

DETAILED DESCRIPTION:
Aim :asseing the effect of intraligmentary dexamethasone on anesthetic efficacy of inferior alveolar nerve block and buccal infiltratation in lower first molar with irreversible pulpitis and apical periodontits, dexamethasone has antiinflammatory effect so it will improve the efficacy of anathesia and reduce postoperative by inhibition the production of phosopholipase and reduction of prostaglandins synthesis

Methods: diagnose the case clinically and readiographically Patients will divide into 3 groups First group will be given inferior alveolar nerve block 4%articaine Hcl1:100 epinephrine Second group will be given inferior alveolar nerve block 4%articaine with intraligmentary dexamethasone Third group will be given buccal infiltratation 4%articaine with intraligmentary dexamethasone After anathesia ,make access cavity and reduce the occulsa surface and make it out of occulsion .

Working length determination will be done by apex locator and confirm it by x ray .

Mechanical preparation will be done by FANTA files and apply EDTA on files Irrigate the canal by Naocl 2.5٪ Complete the root canal preparation through single visit. Obturate the canal by single cone technique and bioceramic sealer. During procedures , record pain intensity on HP visual scale Follow up the patient after 6,12,24 and 48 hours Describe Ibuprofen 200mg in case of sever pain Conclusion : it's predictable that the intraligmentary dexamethasone will reduce the pain during and after root canal procedures

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-45 years old.
2. Systemically healthy patient (ASA I or II).
3. Lower first molar with:

   * Preoperative sharp pain.
   * Slight widening in the periodontal ligament (PDL).
   * Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).

Exclusion Criteria:

1. Patients allergic to anesthetics, or dexamethasone (other corticosteroids).
2. Pregnant or nursing females.
3. Patients having significant systemic disorder (ASA III or IV).
4. Hemostatic disorders or anti-coagulant therapy during the last month.
5. Consumption of opioid or non-opioid analgesics or corticosteroids during the last 12 h before treatment.
6. Retreatment cases.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain | During procedure
  Efficacy of buccal infiltration anesthesia and inferior alveolar nerve block measured during procedures of root canal treatment using numerical rating scale.It is a line numbered from 0-10 , where pain levels are categorized as follows: 0= no pain, 1-3 = mild pain, 4-6= moderate pain, 7-10= severe pain, "10" being the most intense pain conceivable.And instruct patient to raise his hand if he feels pain to reasse if he needs supplementary anathesia

SECONDARY OUTCOMES:
Post-operative pain | After procedure until 48hour
  Patient will record the pain on numerical rating scale (6,12,24 &48h)..It is a line numbered from 0-10 , where pain levels are categorized as follows: 0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10 = severe pain, "10" being the most intense pain conceivable
Number of needed analgesic tablets in case of intolerable pain | After procedure until 48hour
  Ibuprofen 200mgm tabs have been described to patient in case of sever pain (above6)

CONTACTS AND LOCATIONS:
Overall Officials: Angie G Ghoneim, Study Director — Faculty of oral and dental medicine,Cairo university

IPD SHARING:
Plan to Share IPD: No